CLINICAL TRIAL: NCT01198236
Title: Efficacy of Itraconazole as Secondary Prophylaxis in Patients Undergoing Allogeneic Stem Cell Transplantation or Chemotherapy With Prior Invasive Fungal Infection
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Zhejiang University (Other)
Collaborators: Shanghai General Hospital, Shanghai Jiao Tong University School of Medicine (Other); Zhejiang Provincial Hospital of TCM (Other); First Affiliated Hospital of Wenzhou Medical University (Other); Guangdong Provincial People's Hospital (Other)
Responsible Party: Shushen Zheng, The president of the Hospital, The First Hospital of Zhejiang Medical Colleage, Zhejiang University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: SpoIV-CHA-IIS-0802; ITRFUN4044 (Other Grant/Funding Number: Xi'an-Janssen pharmaceutical Ltd.)
Record Dates: First submitted 2010-09-09; First posted 2010-09-10 (Estimated); Last update posted 2011-10-14 (Estimated); Status verified 2011-10

CONDITIONS: Invasive Fungal Infection
Keywords: hematological malignancy; previous proven or probable invasive fungal infection
MeSH Terms: conditions — Invasive Fungal Infections; Hematologic Neoplasms | interventions — Itraconazole; Solutions

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Drug: Itraconazole — Itraconazole will be administered intravenously 2×200 mg/d(200mg twice a day, with 12 hours interval, and should be completed in no less than 60 minutes each time) in the first two days of treatment as a loading dose, then 200mg/d intravenously (200mg once a day with 24 hours interval and completed in no less than 60 minutes) until the end of the at-risk period.
  In transplant patients, the end of "at-risk period" is defined as a stable engraftment of 1*109/L neutrophil cells; in patients who have undergone chemotherapy, it is defined as the resolution of neutropenia (neutrophil cells> 0.5*109/L).
  If needed, the patients will take itraconazole solution orally after intravenous administration.
  Other Names: Sporanox IV and Oral solution

SUMMARY:
Invasive fungal infections (IFI) remain the major cause of death among neutropenic patients receiving chemotherapy for leukemia, or submitted to stem cell transplantation. Patients with a history of invasive fungal infection (IFI) are at high risk of developing relapse and fatal complications.

Prompt intensive antifungal therapy, have improved responses and survival, allowing an increase of antifungal treatments, including secondary antifungal prophylaxis.

Few studies have addressed the role of previous IFI in the feasibility of stem cell transplant, or the secondary prophylaxis with antifungal drugs in preventing recurrence of infection after transplantation. However, given the lack of prospective studies, the role of secondary antifungal prophylaxis remains unclear.

Itraconazole is a wide-spectrum triazole antifungal agent active against Candida albicans, non-albicans, Aspergillus spp., Blastomyces dermatitidis, Blastomyces coccidioides, Cryptococcus neoformans, Sporothrix schenkii, Paracoccidioides brasiliensis, Histoplasma spp. and various kinds of yeast fungi and mycetes.

The role of itraconazole IFI prophylaxis treatment has been proved by many interventional studies. In this prospective, multicentric study of secondary prophylaxis, itraconazole will be given at standard dose to patients undergoing allogeneic stem cell transplantation or chemotherapy with prior invasive fungal infection, to assess the efficacy and safety of itraconazole secondary prophylaxis.

ELIGIBILITY:
Inclusion Criteria:

* Man or woman between 18 and 65 years of age, inclusive.
* Patients who affected by hematological malignancies, receiving chemotherapy, or submitted to stem cell transplantation.
* Patients with previous proven or probable invasive fungal infections, with residual or absent lesions on CT scan or X-ray and the absence of clinical signs of fungal infection at the time of enrollment. Or, possible IFI patients without microbiological evidence but with effective anti-fungal therapy history.

(The diagnosis is according to the definitions of Chinese guideline for the diagnosis and treatment of invasive fungal infections in immunocompromised patients with cancer cancer and hematopoietic stem cell transplant.)

* Subjects (or their legally acceptable representatives) must have signed an informed consent document indicating that they understand the purpose of and procedures required for the study and are willing to participate in the study.
* Lack of clinical symptoms of invasive fungal infection

Exclusion Criteria:

* Patient has no response to the previous intravenous itraconazole antifungal therapy.
* Currently taking the contra-indicated medications such as teldane, astemizol, cisapride and HMG-CoA reductase inhibitor（e.g. Simvastatin, ovastatin, oral Midazolam and Triazolam）
* History of allergy or intolerance to imidazole or azoles anti-fungal agents（e.g. Fluconazol, Itraconazole, Ketoconazole, Miconazole, Clotrimazole）
* Pregnant women, lactating women or women of child bearing potential without applying valid contraceptive measures
* Patients with current cardiac dysfunction (especially with congestive heart failure) or with the history of congestive heart failure
* Patients with severe liver dysfunction (aminotransferase levels ≥5 times the upper limit of normal and total bilirubin level ≥3mg/dL(51.3 μmol/L); or the severity of liver dysfunction does not match this criteria but the patient is in bad condition and not suitable for this trial( doctors make the decision);
* Patients with renal insufficiency having serum Ccr level <30ml/min, calculated from the following formula:

Male: Ccr (ml/min)=(140-age)×weight (kg) /(0.8136×Crea (μmol/L) ) Female:Ccr (ml/min)=(140-age)×weight (kg) ×0.85/(0.8136× Crea (μmol/L) )

* Patients received any experimental drug within 10 days before the planned start of treatment.
* Patients with bad whole body status and not suitable for the trial (doctors make the decision)

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 150 (Actual)
Dates: Start 2008-07; Primary Completion 2010-09 (Actual); Study Completion 2010-11 (Actual)

PRIMARY OUTCOMES:
successful prophylaxis rate | more than 7 days
  The rate of patients without documented relapse of the fungal infection and the absence of new proven, probable or possible IFI at the end of secondary prophylaxis treatment and 7 days later.

SECONDARY OUTCOMES:
rate of patients who developed persistent fever or pulmonary infiltrates of unknown etiology | at least 7 days
  The rate of patients who developed persistent fever or pulmonary infiltrates of unknown etiology. For those neutropenic patients with persistent fever, antibiotics should be used according to the International anti-infection guideline in order to exclude the possibility of bacterial infection. If the fever persists after 5-6 days' combination use of itraconazole and antibiotics, this case would be regarded as "secondary prophylaxis failure" and the trial is terminated , while doctors should search for further clinical therapy to save the patient.

CONTACTS AND LOCATIONS:
Overall Officials: He Huang, MD, Principal Investigator — The First Hopspital of Zhejiang Medical Colleage, Zhejiang University
Locations (1):
- The First Hospital of Zhejiang Medical Colleage Zhejiang University, Hangzhou, Zhejiang, China

REFERENCES:
- [Background] Cordonnier C, Maury S, Pautas C, Bastie JN, Chehata S, Castaigne S, Kuentz M, Bretagne S, Ribaud P. Secondary antifungal prophylaxis with voriconazole to adhere to scheduled treatment in leukemic patients and stem cell transplant recipients. Bone Marrow Transplant. 2004 May;33(9):943-8. doi: 10.1038/sj.bmt.1704469. PMID 15034546
- [Background] de Fabritiis P, Spagnoli A, Di Bartolomeo P, Locasciulli A, Cudillo L, Milone G, Busca A, Picardi A, Scime R, Bonini A, Cupelli L, Chiusolo P, Olivieri A, Santarone S, Poidomani M, Fallani S, Novelli A, Majolino I. Efficacy of caspofungin as secondary prophylaxis in patients undergoing allogeneic stem cell transplantation with prior pulmonary and/or systemic fungal infection. Bone Marrow Transplant. 2007 Aug;40(3):245-9. doi: 10.1038/sj.bmt.1705720. Epub 2007 May 28. PMID 17529996